CLINICAL TRIAL: NCT06015230
Title: A Phase Ⅰb/Ⅱ, Randomized, Double-blind, Placebo-controlled Study to Investigate the Tolerability, Safety,Pharmacokinetics and Efficacy of an Intravenous Treatment Regimen of GR1603 in Subjects with Systemic Lupus Erythematosus
Brief Title: Clinical Study to Investigate the Safety, Tolerability, and Pharmacokinetics of GR1603 in SLE
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR1603-002
Record Dates: First submitted 2023-06-01; First posted 2023-08-29 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: IFNR; Autoimmune Diseases; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Treatment group 1-Ⅰb (Experimental): 6 subjects in GR1603 low dose，2 subjects in placebo
  Interventions: Biological: low dose GR1603 in phase Ⅰb
- Treatment group 2-Ⅰb (Experimental): 6 subjects in GR1603 high dose，2 subjects in placebo
  Interventions: Biological: high dose GR1603 in phaseⅠb
- treatment group 3-Ⅱ (Experimental): low dose GR1603 monthly
  Interventions: Biological: low dose GR1603 in phase Ⅱ
- treatment group 4-Ⅱ (Experimental): high dose GR1603 monthly
  Interventions: Biological: high dose GR1603 in phase Ⅱ
- treatment group 5-Ⅱ (Placebo Comparator): placebo
  Interventions: Biological: Placebo in phase Ⅱ

INTERVENTIONS:
Biological: low dose GR1603 in phase Ⅰb — 6 subjects in GR1603 low dose，2 subjects in placebo
  Arms: Treatment group 1-Ⅰb
Biological: high dose GR1603 in phaseⅠb — 6 subjects in GR1603 high dose，2 subjects in placebo
  Arms: Treatment group 2-Ⅰb
Biological: low dose GR1603 in phase Ⅱ — low dose GR1603 monthly
  Arms: treatment group 3-Ⅱ
Biological: high dose GR1603 in phase Ⅱ — high dose GR1603 monthly
  Arms: treatment group 4-Ⅱ
Biological: Placebo in phase Ⅱ — Placebo
  Arms: treatment group 5-Ⅱ

SUMMARY:
A Study to Investigate the Tolerability, Safety,Pharmacokinetics and efficacy of GR1603 in subjects with Systemic Lupus Erythematosus ； GR1603 injection is a monoclonal antibody targeting IFNAR1, which can block IFNAR binding to type I interferons such as IFNα and be used to treat systemic lupus erythematosus.

DETAILED DESCRIPTION:
This is a Phase Ib/Ⅱ,double blind, multiple-dose study to evaluate the pharmacokinetics (PK), safety，tolerability and efficacy of intravenously administered GR1603 in participants with active SLE despite receiving standard of care .

Phase Ib is a multi-dose escalation phase in which 16 subjects are scheduled to enroll.

A total of 120 subjects were randomly assigned to GR1603 injection low dose group, high dose group or placebo group in phase Ⅱ.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE according to the ACR 1997 ≥24 weeks
* Active moderate to severe SLE
* At least one of these antibodies positive: ANA, anti-dsDNA and anti-Smith.

Exclusion Criteria:

* Active severe or unstable neuropsychiatric SLE
* Clinically significant laboratory test
* Clinically significant active infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2028-06-10 (Estimated); Study Completion 2028-10-04 (Estimated)

PRIMARY OUTCOMES:
Adverse events(phase Ib) | up to week 16
  to characterise the safety and tolerability of GR1603,including abnormal vital signs,laboratory tests,electrocardiogram and physical examination
Number of participants who achieved BICLA response (phase Ⅱ) | week 24
  BICLA respnse:reduction of all baseline BILAG-2004 A to B/C/D and baseline BILAG-2004 B to C/D, and no BILAG-2004 worsening in other organ systems, as defined by ≥1 new BILAG-2004 A or ≥2 new BILAG-2004 B

SECONDARY OUTCOMES:
Cmax(phaseⅠb） | up to week 16
  Pharmacokinetic indices
AUC0-t(phaseⅠb） | up to week 16
  Pharmacokinetic indices
AUC0-∞(phaseⅠb） | up to week 16
  Pharmacokinetic indices
AUCss(phaseⅠb） | up to week 16
  Pharmacokinetic indices
Tmax(phaseⅠb） | up to week 16
  Pharmacokinetic indices
t1/2z(phaseⅠb） | up to week 16
  Pharmacokinetic indices
Vz(phaseⅠb） | up to week 16
  Pharmacokinetic indices
CLz(phaseⅠb） | up to week 16
  Pharmacokinetic indices
Number of participants who achieved SRI (4)(phase Ⅱ) | up to week 28
  An SRI (4) responder defined as a participant who had a reduction in baseline Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score of greater than or equal to 4 points;
Number of participants who achieved BICLA response(phase Ⅱ) | up to week 28
  BICLA respnse:reduction of all baseline BILAG-2004 A to B/C/D and baseline BILAG-2004 B to C/D, and no BILAG-2004 worsening in other organ systems, as defined by ≥1 new BILAG-2004 A or ≥2 new BILAG-2004 B
Number of participants with a ≥50% reduction in CLASI activity score (phase Ⅱ) | up to week 28
  CLASI:Cutaneous Lupus Erythematosus Disease Area and Severity Index
Flare rate(phase Ⅱ） | up to week 28
  A flare was defined as either 1 or more new BILAG-2004 A or 2 or more new BILAG-2004 B items compared to the previous visit

CONTACTS AND LOCATIONS:
Overall Officials: xiaofeng zeng, PHD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking union Medical Hosipital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No